CLINICAL TRIAL: NCT04857515
Title: An Exploratory, Observational, Open-label, Remote Study of Clickotine: A Digital Therapeutic
Brief Title: Clinical Learning Study for a Mobile Smoking Cessation Program
Status: Completed | Type: Observational
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-101-CLS-001
Record Dates: First submitted 2021-04-01; First posted 2021-04-23 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation; Smoking Behaviors; Smoking Reduction; Smoking, Cigarette; Smoking; Nicotine Dependence
Keywords: Smoking Cessation; Smoking Cessation Program; Smoking Cessation Digital Therapeutic
MeSH Terms: conditions — Smoking Cessation; Smoking; Smoking Reduction; Cigarette Smoking; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cigarette Smokers: Adult cigarette smokers who only smoke combustible cigarettes
  Interventions: Device: Clickotine®
- Dual-Users: Adult smokers who smoke both combustible cigarettes and vape
  Interventions: Device: Clickotine®

INTERVENTIONS:
Device: Clickotine® — Clickotine is a DTx that contains behavior modification techniques that include controlled breathing, social engagement, personalized messaging, medication access and adherence, digital diversions, and financial incentives.

SUMMARY:
The purpose of this study are to obtain learnings regarding the Digital Therapeutic (DTx) experience of Clickotine, including acceptability and preference of the overall program and specific DTx components, as well as to obtain learnings related to adult participants' use of the DTx for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age 18 and older.
* For cigarette smokers: Smokes at least 5 cigarettes a day. For dual-users: Smokes cigarettes AND uses e-cigarettes, with the following additional criteria:

  * Smokes at least 5 cigarettes a day
  * Vaping sessions, when they occur, must be for at least 10 minutes (15 puffs)
* Fluent in written and spoken English (confirmed by ability to read and comprehend the informed consent form)
* Lives in the United States.
* Is the solo user of an iPhone with iPhone operating system (iOS)13 or greater capabilities or a smart phone with an Android operating system (OS) 9 or greater capabilities.
* Has an active email address.
* Willing and able to receive SMS text messages on their smartphone and email messages.
* Have access to internet connection during the study duration.
* Able to confirm download of installed DTx on baseline date.
* Willing and able to comply with study protocol and assessments.
* Is willing and able to self-identify sessions of cigarette smoking (1 or more consecutive cigarettes) or vaping (approximately 15 puffs or around 10 minutes in duration) and log those sessions.
* Self-reported comfort with and ability to use smartphone apps/programs.

Exclusion Criteria:

* Prior use of Clickotine.
* Currently using a software app for smoking cessation.
* Lifetime diagnosis of schizophrenia, psychotic disorder, or pervasive developmental disorders, as per participant self-report.
* Any unstable medical illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrine, neurologic (including history of severe head injury with loss of consciousness), immunologic, or hematologic disease, as per participant self-report.
* Other significant medical condition that, in the opinion of the Investigator or study sponsor, may cofound the interpretation of device efficacy, safety, and tolerability.
* Current use of tobacco-containing products other than cigarettes or e-cigarettes (e.g. snuff, chewing tobacco, cigars, or pipes).
* Does not have or is unwilling to create a PayPal account

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age: 18+ US Resident Fluent in english
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
The main outcome of the Clickotine Learning Study is to determine acceptability of the digital intervention (DTx). | 4 Months
  General acceptability of the DTx will be evaluated via surveys for all participants
The main outcome of the Clickotine Learning Study is to determine engagement with the digital intervention (DTx). | 4 Months
  Engagement with the digital intervention will be measured via app use for all participants
The main outcome of the Clickotine Learning Study is to evaluate attitudes and beliefs regarding the digital intervention. | 4 Months
  Attitudes and beliefs regarding the digital intervention will be evaluated by interview for selected participants

SECONDARY OUTCOMES:
The secondary outcome of the Clickotine Learning Study is to measure engagement levels with the digital intervention for cigarette smokers as compared to dual-users | 4 Months
  These engagement levels will be measured via app use.
The secondary outcome of the Clickotine Learning Study is to determine acceptability of the digital intervention for cigarette users as compared to dual-users | 4 Months
  Acceptability of the digital intervention will be evaluated via survey

CONTACTS AND LOCATIONS:
Locations (1):
- Click Therapeutics, New York, New York, United States